CLINICAL TRIAL: NCT00798005
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Efficacy and Safety Study of Different Doses and Schedules of Administration of NV1FGF in Patients With Severe Peripheral Artery Occlusive Disease.
Brief Title: Efficacy and Safety Study of NV1FGF in Patients With Severe Peripheral Artery Occlusive Disease.
Acronym: TALISMAN202
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI6144; NV1FGF-PM202
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Severe Peripheral Artery Occlusive Disease
Keywords: NV1FGF; PAOD; CLI
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: XRP0038 (NV1FGF)

SUMMARY:
Peripheral Arterial Occlusive Disease (PAOD) is a condition caused by ischemia in the legs due to atherosclerotic disease affecting the larger arteries of the legs. Chronic PAOD can be regarded as a marker of generalized atherosclerosis. PAOD threatens the survival of an extremity and often causes lifelong disablement from a painful leg. The clinical consequences of PAOD include pain on walking (claudication), pain at rest and loss of tissue integrity in the distal limbs.A variety of medical therapies have been investigated for patients with PAOD. There is currently no evidence to suggest that any medical therapy is effective for patients with rest pain and/or ischemic ulcers.

Also, the use of intramuscular angiogenic VEGF-A gene transfer has recently demonstrated a improvement in clinical and hemodynamic status in patients with severe PAOD

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent was to be signed before proceeding with any study procedure.
2. Patients with severe PAD.
3. Trophic lesions with no signs of healing (no reduction in ulcer size or depth) for at least 2 weeks prior to first study treatment administration (Day 1).
4. Patients with objective evidence of peripheral vascular disease in the diseased limb on 2 consecutive examinations performed at least 1 week apart.
5. Demonstration or documentation of total occlusion of the affected limb of one or more of the iliac, superficial femoral, popliteal and/or one or more infrapopliteal arteries as assessed by angiography or magnetic resonance angiography (MRA)
6. Transcutaneous oxygen pressure (TcPO2): mean resting supine TcPO2 of the foot of ≤40 mmHg based on 2 separate measures performed at least 1 week apart
7. Poor/not candidates for revascularization

Exclusion criteria

1. Previous or current history of malignant disease.
2. Positive cancer screening (liver, prostate, colon, cervix, breast, lung)
3. Successful lower extremity surgery (bypass/angioplasty of the leg to be treated) within 3 months prior to the first administration of study treatment [Day 1]).
4. Patients planned to undergo amputation of target limb within 1 month following the first administration of study treatment.
5. Patients with a history of severe renal failure.
6. Creatinine >2.0 mg/dL (176 µmol/L) or estimated creatinine clearance <30 mL.
7. Serious concomitant medical conditions not adequately controlled (other than severe PAD),
8. Buerger's disease.
9. Patients in dialysis.
10. Active proliferative retinopathy
11. Patients who had a stroke or neurologic deficit presumed to be due to stroke within 3 months prior to the first administration of study treatment.
12. Previous treatment with any angiogenic growth factor.
13. Positive serology for HIV 1 or 2.
14. Participation in clinical trials of non-approved experimental agents within 4 weeks before study entry.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2002-06; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
evaluate the efficacy and the safety of NV1FGF compared to placebo in patients with severe PAOD.

SECONDARY OUTCOMES:
evaluate the biodistribution of NV1FGF and to measure serum levels of antibodies against FGF-1

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

REFERENCES:
- [Result] Henry TD, Mendelsohn F, Comerota A, Pham E, Grek V, Coleman M, Meyer F, Annex B Dose and regimen effects of intramuscular NV1FGF in patients with critical limb ischemia: A randomized, double-blind, placebo controlled study. Eur H J 2006, 27 Suppl 1 Abs P1497
- [Derived] Niebuhr A, Henry T, Goldman J, Baumgartner I, van Belle E, Gerss J, Hirsch AT, Nikol S. Long-term safety of intramuscular gene transfer of non-viral FGF1 for peripheral artery disease. Gene Ther. 2012 Mar;19(3):264-70. doi: 10.1038/gt.2011.85. Epub 2011 Jun 30. PMID 21716303
- See also: Related Info — http://www.sanofi-aventis.com